CLINICAL TRIAL: NCT03877809
Title: A Personalized Medicine Approach for Beta-thalassemia Transfusion Dependent Patients: Testing SIROLIMUS in a First Pilot Clinical Trial
Brief Title: Testing SIROLIMUS in Beta-thalassemia Transfusion Dependent Patients
Acronym: SIRTHALACLIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rare Partners srl Impresa Sociale (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT2-02-17; 2018-001942-33 (EudraCT Number); 208872/Z/17/Z (Other Grant/Funding Number: Wellcome Trust (Innovator Award))
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Beta-Thalassemia
Keywords: Fetal hemoglobin; Sirolimus; Red Blood Cells
MeSH Terms: conditions — beta-Thalassemia | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Interventional, pilot, single centre, open-label phase II study with sirolimus in patients with transfusion dependent beta-thalassemia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label trial (Experimental): Sirolimus 0.5 mg tablets
  Interventions: Drug: Sirolimus 0.5 mg

INTERVENTIONS:
Drug: Sirolimus 0.5 mg — Daily administration of 1 or more tablets

SUMMARY:
Beta-thalassemias are hereditary blood disorders caused by reduced or absent synthesis of hemoglobin beta chains, with variable outcomes ranging from severe anemia to clinically asymptomatic individuals. Treatment is symptomatic and thalassemia is a major unmet medical need. Survival is increased, even in patients needing transfusions, in comparison with a few years ago, but the quality of life is poor for many patients. In some patients, an anomalous expression of gamma-globin genes has been observed, with a consequent rise in Fetal Hemoglobin levels. The patients displaying a clinical phenotype known as Hereditary Persistence of Fetal Hemoglobin (HPFH) exhibit a positive clinical status. To mimick HPFH, several compounds able to induce expression of fetal hemoglobins (HbF) have been evaluated. Within this framework, sirolimus is particularly interesting as an inducer of HbF. It has been used for many years for different indications and the available preclinical evidence warrant the start of a clinical development plan in thalassemia. The investigators propose a clinical trial in beta-thalassemia patients, designed to evaluate the effect of sirolimus on several parameters related to red blood cell status and to the level of HbF in particular, as a first step for the full clinical development in this new indication.

DETAILED DESCRIPTION:
The general aim of the protocol is to demonstrate the applicability of a personalised and precision medicine approach in beta-thalassemia in a clinical trial setting for a repurposed drug, namely sirolimus. The presence of high level of Fetal Hemoglobin (HbF) is considered a condition predictive of a favourable outcome in thalassemia and its increase induced by pharmacological agents is considered a potential way to improve clinical status of the patients. In the present trial, in terms of efficacy analysis, the investigators will focus their attention on HbF levels.

Primary objective:

• To evaluate the suitability of sirolimus for the treatment of beta-thalassemia patients within the frame of a comprehensive project aimed to the reduction of their transfusions need (consequently ameliorating their quality of life). This goal can be obtained through a pharmacologically mediated increased level of HbF, with a prerequisite to be verified, namely the correlation between induction of HbF in vitro and in vivo in single patients.

Secondary objectives:

* To assess safety of sirolimus and correlation between administered dose and blood levels in beta-thalassemia patients,
* To assess the influence of sirolimus on transfusion regimen
* To assess the effect of sirolimus on hematopoietic and immune system of thalassemia patients.

ELIGIBILITY:
* Patients over 18 years of age;
* Patient able to understand the informed consent and to sign it before any study procedure;
* With β+/β+ and β+/β0 thalassemia genotype;
* Documented diagnosis of major or intermediate thalassemia transfusion-dependent (nr of transfusion not less than 8 over the past 12 months before selection);
* On regular transfusion since at least 6 years;
* With splenectomy performed at least 60 days before selection or spleen dimensions < 20 cm in the largest part as detected by abdominal echography;
* Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years or female participants of childbearing potential using and/or willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or using any other method considered sufficiently reliable by the investigator in individual cases. Patients must be counseled concerning measures to be used to prevent pregnancy and potential toxicities prior to the first dose of sirolimus;
* Patient willing to follow all the study requirements and perform all the study visits and to cooperate with the investigator;
* Patient followed by the same clinical site since at least 6 months.

Note that patients will be treated with oral sirolimus only in the case their Erythroid Precursor Cells (ErPCs) are responsive to the in vitro treatment with sirolimus according to laboratory specific definition (≥ 20% increase of HbF in comparison with samples not treated with sirolimus);

Exclusion Criteria:

* Patient treated with hydroxyurea at selection visit or in the last 6 months;
* Ongoing treatment with drugs possibly affecting sirolimus actions;
* Documented aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x Upper Limit of Normal (ULN) at selection;
* Documented Platelet count <150.000/microliter and >1.000.000/microliter at selection;
* Heart failure as classified by the New York Heart Association (NYHA) classification 3 or higher;
* Uncontrolled hypertension defined as systolic blood pressure (BP) ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg;
* Significant arrhythmia requiring treatment,
* Corrected QT interval> 450 msec on selection ECG;
* Ejection fraction <50% by echocardiogram, multiple gated acquisition scan or cardiac magnetic resonance;
* Myocardial infarction within 6 months prior of selection;
* Positivity for human immunodeficiency virus (HIV) antibody, active hepatitis B (HBV) or hepatitis C (HCV) as demonstrated by the presence of hepatitis B surface antigen (HBsAg) and a positive HCV-RNA test, HBcAb and HBV-DNA positivity
* White blood cell [WBC] count <3000 cells per μL and/or Granulocytes <1500/mm3;
* Total cholesterol > 240 mg/dl;
* Triglycerides > 200 mg/dl;
* Proteinuria with urinary protein >1g/24 hrs;
* Current participation in another trial with investigational drug or experimental device, or inclusion in another trial with investigational drug or experimental device within the preceding month;
* Major surgery (including splenectomy) within 60 days before selection (patients must have fully recovered from any previous surgery);
* Iron chelation therapy changed in the last 3 months prior to selection (note that Deferiprone is not accepted as a chelation therapy drug in this study while Desferioxamine and Deferasirox are tolerated at stable dose);
* Current treatment with macrolide antibiotics (clarithromycin);
* Pregnant or lactating women;
* History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the experimental drug;
* Treatment with live vaccines within 90 days preceding the selection;
* Subject with history or current malignancies (solid tumors and haematological malignancies) or presence of masses/tumor detected by ultrasound at selection;
* Subject with any significant medical condition and/or laboratory abnormality considered by the investigator as not adequately controlled at the time of selection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of fetal hemoglobin level | 360 days
  Fetal hemoglobin level in peripheral blood at day 360 compared to day 0, assessed through high pressure liquid chromatography (HPLC)

SECONDARY OUTCOMES:
Change from baseline of fetal hemoglobin level | 180 days
  Fetal hemoglobin level in peripheral blood at days 90 and 180 compared to day 0, assessed through HPLC
Change from baseline of γ-globin expression | 360 days
  Level of induction of the γ-globin expression at day 90, 180 and 360 compared to day 0
Change from baseline of biomarkers for erythropoiesis | 360 days
  - - Evaluation of the biomarkers for erythropoiesis level at day 180 and 360 compared to baseline. Biomarkers will include: Reticulocytes count, Nucleated red blood cells count
Change from baseline of biomarkers for erythropoiesis | 360 days
  - - Evaluation of the biomarkers for erythropoiesis level at day 180 and 360 compared to baseline. Biomarkers will include: erythropoietin level, serum transferrin receptor level.
Change from baseline of biomarkers for haemolysis | 360 days
  - Evaluation of the biomarkers for haemolysis level at day 180 and 360 compared to baseline. Biomarkers will include: serum bilirubin level
Change from baseline of biomarkers for haemolysis | 360 days
  - Evaluation of the biomarkers for haemolysis level at day 180 and 360 compared to baseline. Biomarkers will include: serum lactate dehydrogenase (LDH) level
Change from baseline of tranfusion needs | 360 days
  - Measurement of the total blood quantity (in mL) transfused and recording of the number of transfusions done in a semester (day -360 to -180, day -180 to 0, day 0 to 180, day 180 to 360)
Change from baseline of Iron status | 360 days
  * Evaluation of the intake of iron chelators at days 180 and 360 compared to baseline
  * Evaluation of serum ferritin level at day 90, 180 and 360 in comparison with day 0
Change from baseline of Immune function | 360 days
  * Peripheral blood immunophenotype-Lymphocyte subsets at day 90 and 360 compared to day 0
  * Quantitative analysis of ImmunoglobulinG/ImmunoglobulinA/ImunoglobulinM at day 90 and 360 compared to day 0
Change from baseline of Quality of Life | 360 days
  Evaluation of the patient quality of life at 6 and 12 months compared to baseline through Transfusion-dependent Quality of Life questionnaire (TranQol), measuring specifically the quality of life in patients with thalassemia. The TranQol is a disease-specific Quality of Life measure that has been shown to be valid and reliable (Klaassen et al, British Journal of Haematology, 2014, 164, 431-437). On a total scale of 0-100, higher values always represent a better outcome. The questions are grouped into four domains: physical health, emotional health, family functioning, and school and career functioning. The adult self-report questionnaires include a fifth category on sexual activity which is only one item. Subscales are summed.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Department of Life Sciences and Biotechnology, Section of Biochemistry and Molecular Biology, Ferrara
  - Department of Growth and Reproduction Azienda Ospedaliero-Universitaria S.Anna, Ferrara

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study the study protocol and the clinical trial report will be available to other researchers. Publication of the data is planned
Supporting Information: Study Protocol, CSR
Time Frame: After completion of the Clinical Study Report preparation
Access Criteria: Free availability of the publication. Free availability of the study protocol upon request

REFERENCES:
- [Result] Zuccato C, Cosenza LC, Zurlo M, Gasparello J, Papi C, D'Aversa E, Breveglieri G, Lampronti I, Finotti A, Borgatti M, Scapoli C, Stievano A, Fortini M, Ramazzotti E, Marchetti N, Prosdocimi M, Gamberini MR, Gambari R. Expression of gamma-globin genes in beta-thalassemia patients treated with sirolimus: results from a pilot clinical trial (Sirthalaclin). Ther Adv Hematol. 2022 Jun 21;13:20406207221100648. doi: 10.1177/20406207221100648. eCollection 2022. PMID 35755297
- [Derived] Zurlo M, Finotti A, Gamberini MR, Gambari R. Co-Induction of ULK-1 and AHSP mRNAs in Erythroid Precursor Cells Isolated From a Sirolimus-Treated beta-Thalassemia Patient: A Case Report Study. Br J Biomed Sci. 2025 Jun 27;82:14311. doi: 10.3389/bjbs.2025.14311. eCollection 2025. PMID 40655320
- [Derived] Zurlo M, Nicoli F, Proietto D, Dallan B, Zuccato C, Cosenza LC, Gasparello J, Papi C, d'Aversa E, Borgatti M, Scapoli C, Finotti A, Gambari R. Effects of Sirolimus treatment on patients with beta-Thalassemia: Lymphocyte immunophenotype and biological activity of memory CD4+ and CD8+ T cells. J Cell Mol Med. 2023 Feb;27(3):353-364. doi: 10.1111/jcmm.17655. Epub 2023 Jan 10. PMID 36625233